CLINICAL TRIAL: NCT00663182
Title: Entecavir for Patients With Decompensated HBV-Related Cirrhosis:a Prospective Randomized Controlled Trial
Brief Title: Entecavir for Patients With Decompensated Hepatitis B Virus (HBV)-Related Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Jian Shi, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Entecavir-01
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Hepatitis B Virus; Decompensated Cirrhosis
Keywords: Entecavir; cirrhosis; anti-viral; therapy
MeSH Terms: conditions — Hepatitis B; Fibrosis | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients with decompensated HBV-related cirrhosis
  Interventions: Drug: Entecavir
- B (No Intervention): Untreated

INTERVENTIONS:
Drug: Entecavir — Entecavir 0.5 mg/d
  Other Names: Baraclude
  Arms: A

SUMMARY:
The aim of this study is to evaluate the effect of Entecavir for patients With decompensated HBV-Related cirrhosis.

DETAILED DESCRIPTION:
Chronic hepatitis B is one of the most widespread viral infections worldwide, potentially leading to liver cirrhosis and hepatocellular carcinoma. Previous studies demonstrated that patients with active viral replication, defined as the presence of detectable serum HBV-DNA or HBeAg, were at increased risk of developing progressive liver disease or death.The prognosis of decompensated cirrhosis resulting from chronic hepatitis B virus infection is poor. Anti-viral therapy in decompensated HBV-related cirrhosis has been recommended by the American Association for the Study of Liver Diseases. However, no high quality research on the effectiveness of anti-viral therapy in decompensated cirrhosis has been performed.

Entecavir is a new nucleotide analogue, which has been proved effective in suppressing viral replication and decreasing the necroinflammatory response, was recommended as a first-line medication in AASLD guideline. Our purpose was to evaluate the effect of Entecavir for patients With decompensated HBV-Related cirrhosis. The main outcomes were liver function, HBV-DNA, disease progression, hepatocellular carcinoma, Child-Pugh score and the survival.

ELIGIBILITY:
Inclusion Criteria:

1. over 16 years of age;
2. evidence of active viral replication was documented by a positive test for HBV-DNA in serum;
3. Liver cirrhosis was proven by ultrasound or CT;
4. Decompensated cirrhosis was evidenced by a Child-Pugh score ≥ 7;
5. patients had decompensation signs such as jaundice, ascites, variceal bleeding, hepatic encephalopathy

Exclusion Criteria:

1. evidence of hepatocellular carcinoma (suspicious foci on hepatic ultrasonography at screening or a rising serum level of alpha-fetoprotein)
2. a serum alanine aminotransferase level more than 10 times the upper limit of normal
3. coinfection with hepatitis C or D virus or human immunodeficiency virus
4. other types of cirrhosis
5. a history of anti-viral therapy
6. a total bilirubin level higher than 170 mmol/L
7. a history of malignant tumors

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
liver function | 1 year
HBV-DNA | 1 year

SECONDARY OUTCOMES:
disease progression | 2 years
hepatocellular carcinoma | 2 year
Child-Pugh score | 2 year
motality | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Shi, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Result] Tseng PL, Lu SN, Tung HD, Wang JH, Changchien CS, Lee CM. Determinants of early mortality and benefits of lamivudine therapy in patients with hepatitis B virus-related decompensated liver cirrhosis. J Viral Hepat. 2005 Jul;12(4):386-92. doi: 10.1111/j.1365-2893.2005.00608.x. PMID 15985009
- [Result] Villeneuve JP, Condreay LD, Willems B, Pomier-Layrargues G, Fenyves D, Bilodeau M, Leduc R, Peltekian K, Wong F, Margulies M, Heathcote EJ. Lamivudine treatment for decompensated cirrhosis resulting from chronic hepatitis B. Hepatology. 2000 Jan;31(1):207-10. doi: 10.1002/hep.510310130. PMID 10613747